CLINICAL TRIAL: NCT02482454
Title: Phase III Study of Radiofrquency Ablation Combined With Cytokine-induced Killer Cells for the Patients With Cholangiocarcinoma
Brief Title: Radiofrquency Ablation Combined With Cytokine-induced Killer Cells for the Patients With Cholangiocarcinoma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Principal Investigator, peng du, Director of Science and Education Division, The First People's Hospital of Changzhou
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: chol001
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-02

CONDITIONS: Cholangiocarcinoma
Keywords: radiofrequency ablation; cytokine-induced killer cells; cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RFA alone (Other): Patients undergo radiofrequency ablation alone.
  Interventions: Procedure: Radiofrequency ablation
- RFA+CIK (Experimental): Autologous cytokine-induced killer cells were transfer via venous one week after RFA
  Interventions: Procedure: Radiofrequency ablation; Biological: Cytokine-induced killer cells

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation is performed percutaneously under CT/US guidance
  Other Names: RFA
Biological: Cytokine-induced killer cells — The patients received autologous cytokine-induced killer cells transfusion one week after RFA treatment.
  Other Names: CIK
  Arms: RFA+CIK

SUMMARY:
The purpose of this study is to determine whether combining of radiofrequency ablation (RFA) and cytokine-induced killer cells (CIK) transfusion can prolong survival of patients with cholangiocarcinoma.

DETAILED DESCRIPTION:
The primary objective is to evaluate whether RFA followed by CIK transfusion can prolong survival of patients with cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed cholangiocarcinoma
* Primary lesions (cholangiocarcinoma) are not resected
* Serum bilirubin level of 2.0 mg/dl or less.
* Performance status of 0 or 1.
* Expected survival of 1 year or more.
* Informed consent from the patient.

Exclusion Criteria:

* With extrahepatic metastases
* With other neoplastic disease that is measurable or being treated other than cholangiocarcinoma.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2030-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 1 year
  Recurrence-free survival (RFS) was defined as the time from the date of RFA to the date of recurrence or the date of the last follow-up.

SECONDARY OUTCOMES:
Adverse events | 4 weeks
  Adverse events related to RFA and CIK treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Changping Wu, M.D., Study Director — The First People's Hospital of Changzhou
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No